CLINICAL TRIAL: NCT00787488
Title: A Pilot Study of Intravenous and Intraperitoneal Chemotherapy Plus Abdominal Hyperthermia to Treat Optimally Debulked and Recurrent Epithelial Ovarian, Fallopian Tube, and Primary Peritoneal Cancers
Brief Title: Pilot Study of IV and IP Chemotherapy Plus Abdominal Hyperthermia for Ovarian Ca
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not funded
Sponsor: Mark Dewhirst (Other)
Responsible Party: Sponsor-Investigator, Mark Dewhirst, Professor, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008510
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Ovarian Cancer
Keywords: Ovarian; debulked; recurrent; Stage III; Stage IV
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Chemotherapy plus Hyperthermia
  Interventions: Device: Hyperthermia

INTERVENTIONS:
Device: Hyperthermia — Every 3 weeks

SUMMARY:
This is a pilot study aimed to test the feasibility and safety of administering combination chemotherapy with paclitaxel (both intravenously and intraperitoneally) and cisplatin (intraperitoneally) plus whole abdominal hyperthermia every 3 weeks in the treatment of optimally debulked, advanced or recurrent ovarian, primary peritoneal, and fallopian tube cancer patients.

DETAILED DESCRIPTION:
Day 1 of each 21 day Cycle:

Paclitaxel 175 mg/m2 IV (infused over 3 hours)

Day 1 or 2 of each Cycle Adequate IV hydration with normal saline (1000 ml recommended)followed by intraperitoneal infusion of 500 ml normal saline through the IP port.

Cisplatin 75 mg/m2 reconstituted in 500 ml NS warmed to 37 degrees Celsius is infused IP (30 minute infusion)followed immediately by whole abdominal hyperthermia

Abdominal hyperthermia will be delivered using the BSD 2000 ellipse system to target temperatures of 40-42 degrees Celsius monitored via rectally and vaginally continuing for no greater than 60 minutes after maximal 30 minute warm-up phase. Total duration of hyperthermia will be no greater than 90 minutes.

Day 8:

Paclitaxel 60 mg/m2 IP. Paclitaxel will be diluted and filtered initially in 1000 ml of normal saline or D5W warmed to 37 degrees Celsius. For IP administration, the patient must receive an additional 1000 ml of normal saline degrees Celsius in the peritoneal cavity.

Cycles will be repeated every 3 weeks x 6 cycles. Patients will be followed until disease progression/recurrence or death.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed Stage III or Stage IV advanced, persistent, or recurrent epithelial ovarian, primary peritoneal, or fallopian tube cancer
* Optimal debulking (< 1cm residual disease) of their disease within 6 weeks of the start of the study
* Patients must have received no more than 2 prior chemotherapy regimens with at least 4 weeks since prior chemotherapy
* GOG performance status 0, 1, or 2
* Patients must have normal organ and marrow function defined as:
* absolute neutrophil count >1,500/mcL
* platelets >100,000/mcL
* total bilirubin and creatinine <1.5 X institutional upper limit of normal(ULN)
* AST(SGOT)/ALT(SGPT)<3 X institutional ULN

Exclusion Criteria:

* Patients with biochemical recurrences or evidence of measurable disease
* Patients with suboptimal (>1 cm) residual disease
* Patients who have had chemotherapy within 4 weeks prior
* Receiving any investigational agents
* Known brain metastases
* Epithelial ovarian carcinoma of low malignant potential (borderline carcinomas)
* Uncontrolled intercurrent illness
* Prior radiation therapy
* History of other invasive or pre-invasive malignancies (except non-melanoma skin cancer) within the past 5 years

Ages: 18 Years to 72 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Toxicity | 6 months

SECONDARY OUTCOMES:
Clinically free of disease. Response definitions will be based on CA-125, clinical assessment, CT imaging | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Jewell, MD, Principal Investigator — Duke University; Angeles Secord, MD, Principal Investigator — Duke University; Ellen Jones, MD, PhD, Principal Investigator — Duke University Medical Center, Radiation Oncology